CLINICAL TRIAL: NCT01668407
Title: Use of a Robot for the Rehabilitation of Walking in Patients With Parkinson's Disease.
Brief Title: Robot Walking Rehabilitation in Parkinson's Disease
Acronym: ROBOPARK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele Roma (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RP 04/12
Record Dates: First submitted 2012-05-08; First posted 2012-08-20 (Estimated); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Idiopathic Parkinson's Disease; Progressive Supranuclear Palsy
Keywords: Parkinson's disease; PSP; Robot; Gait rehabilitation
MeSH Terms: conditions — Parkinson Disease; Supranuclear Palsy, Progressive | interventions — Exercise Test

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Robot-Assisted Gait Training (RAGT) (Experimental): Robot-Assisted Gait Training (RAGT): Subjects (at least 40) will undergo inpatient rehabilitation consisting of a treatment cycle using the GE-O system device, according to individually tailored exercise scheduling. The practice will include robot-assisted walking at variable speeds for 45 min with a partial body weight support (BWS). All participants started with 30-40% BWS and an initial treadmill speed of 1.5 km/h speed will be increased to a range of 2.2 to 2.5 km/h before BWS will be decreased.
  Interventions: Device: Robot-Assisted Gait Training (RAGT)
- Treadmill Gait Training (TT) (Active Comparator): Treadmill Gait Training (TT): Subjects (at least 40) will undergo inpatient rehabilitation consisting of a treatment cycle using the treadmill device, according to individually tailored exercise scheduling. The practice included treadmill walking at variable speed for 45 minutes. All participants will start at an initial treadmill speed of 1.5 km/h speed will be increased to a range of 2.2 to 2.5 km/h.
  Interventions: Procedure: Treadmill Gait Training (TT)

INTERVENTIONS:
Device: Robot-Assisted Gait Training (RAGT) — Subjects (at least 40 subjects) will undergo inpatient rehabilitation consisting of a treatment cycle using the GE-O system device, according to individually tailored exercise scheduling. The practice will include robot-assisted walking at variable speeds for 45 min with a partial body weight support (BWS). All participants started with 30-40% BWS and an initial treadmill speed of 1.5 km/h speed will be increased to a range of 2.2 to 2.5 km/h before BWS will be decreased.
  Other Names: End effector G-EO System
  Arms: Robot-Assisted Gait Training (RAGT)
Procedure: Treadmill Gait Training (TT) — Subjects (at least 40 subjects) will undergo inpatient rehabilitation consisting of a treatment cycle using the treadmill device, according to individually tailored exercise scheduling. The practice included treadmill walking at variable speed for 45 minutes. All participants will start at an initial treadmill speed of 1.5 km/h speed will be increased to a range of 2.2 to 2.5 km/h.
  All the treatment consists of 20 sessions for the lower limbs, each lasting 45 minutes, 5 days a week for 4 weeks.
  Other Names: TREADMILL
  Arms: Treadmill Gait Training (TT)

SUMMARY:
The effectiveness of non-pharmacological treatment on gait impairment on Parkinson Disease (PD) such as exercises has been demonstrated; in particular an example for patient tailored exercises is physiotherapy. The goal of physiotherapy treatment is to enable PD patients to maintain their maximum level of mobility, activity, and independence. Several systematic reviews and clinical studies have shown that physical therapy can contribute to minimize the disabling effects of motor and sensory impairments in order to enhance participation in societal roles and quality of life. The use of electromechanical devices such as treadmill training (a supplement to conventional therapies) in the last years has also been used with PD patients and a systematic Cochrane has been conducted by Mehrholz in 2010 to assess the effectiveness and acceptability of treadmill training in the treatment of gait disorders for patients with PD. In the last years new robotic assisted device can be used in gait training in neurological disorder. Till now only few studies, have focused on the effects of exoskeleton or end effector robot-assisted training in PD patients, with a interesting preliminary results.

DETAILED DESCRIPTION:
The specific aims of this project are:

1. to verify whether the robotics lower limb treatment with body weight support is more effective than the treadmill treatment in the reduction of motor impairment in PD or PSP patients, and to improve the quality of the gait and the endurance;
2. to analyze possible improvements in terms of physiological biomechanical gait through analysis of kinematics , kinetics and EMG evaluation;
3. to analyze possible improvements in terms of reduction of instable posture and movements , which can represent a reduction of the risk of fall typical of these subjects;
4. to evaluate the kinematic, kinetic and EMG quantitative data during selected movements (gait, posture, ) compared with age matched reference data;
5. to investigate the stability of the effects of robot-assisted treatment at 4/6 months follow-up in terms of Quality of Life (QoL).

A first goal of this project is to investigate the differences in improvement of the quality and safety of the gait (motor performance and functional recovery) through kinematic/kinetic and EMG parameters (Change in Step Length, Change in Gait Velocity and Change in Stride Time Variability, 3D joints kinematics, ground reaction forces, joint kinetics, muscle activation,) and traditional clinical scales in Parkinson's patients.

The second goals is aimed at identifying possible advantages in the QoL of patients undergoing such a kind of rehabilitation treatment and at investigating novel methods enabling lower limb functional recovery, leading to wide potential for regaining personal independence.

The third goal is to analyze direct cost savings associated with the use of such technologies, measured as direct, indirect and intangible costs, through specific HTA procedures.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic PD or PSP by UK Brain Bank criteria,
* Age between 18-80;
* Able to walk 25 feet unassisted or with minimal assistance;
* On stable doses of Parkinson's medications for at least 2 weeks prior to study onset;
* Endurance sufficient to stand at least 20 minutes unassisted per patient report.

Exclusion Criteria:

* Other significant neurological or orthopedic problems.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-03-30 (Actual); Primary Completion 2015-08-30 (Actual); Study Completion 2016-03-31 (Actual)

PRIMARY OUTCOMES:
6 minutes walking test. | Change from Baseline in gait speed at 6 months follow up.
  The 6 minuts walking test as primary outcome assessments will be collected 1 hour after oral assumption of levodopa at baseline (inclusion)(T0) and endpoint (after 20 robot session) (T1) (no later than 1 day > last training session) at the follow-up examination after 6 months from the treatments conclusion (T2).

SECONDARY OUTCOMES:
Time Up and Go test. | baseline, weekly during intervention, 6 months follow up.
  Time Up and Go test will be collected 1 hour after oral assumption of levodopa at baseline (inclusion)(T0) and endpoint (after 20 robot session) (T1) (no later than 1 day > last training session) at the follow-up examination after 6 months from the treatments conclusion (T2).
Gait Parameters | baseline, weekly during intervention, 6 months follow up.
  Gait Analysis will be collected 1 hour after oral assumption of levodopa at baseline (inclusion)(T0) and endpoint (after 20 robot session) (T1) (no later than 1 day > last training session) at the follow-up examination after 6 months from the treatments conclusion (T2).

CONTACTS AND LOCATIONS:
Overall Officials: Patrizio Sale, MD, Principal Investigator — IRCCS San Raffale Pisana
Locations (3):
- Italy (3):
  - Polytecnic University of Marche, Ancona
  - San Raffaele Cassino, Cassino
  - IRCCS San Raffaele Pisana, Rome

REFERENCES:
- [Derived] Sale P, Stocchi F, Galafate D, De Pandis MF, Le Pera D, Sova I, Galli M, Foti C, Franceschini M. Effects of robot assisted gait training in progressive supranuclear palsy (PSP): a preliminary report. Front Hum Neurosci. 2014 Apr 17;8:207. doi: 10.3389/fnhum.2014.00207. eCollection 2014. PMID 24860459
- [Derived] Sale P, De Pandis MF, Le Pera D, Sova I, Cimolin V, Ancillao A, Albertini G, Galli M, Stocchi F, Franceschini M. Robot-assisted walking training for individuals with Parkinson's disease: a pilot randomized controlled trial. BMC Neurol. 2013 May 24;13:50. doi: 10.1186/1471-2377-13-50. PMID 23706025